CLINICAL TRIAL: NCT06464835
Title: Effect of ITBS Combined with NMES on Post-stroke Dysphagia and Corresponding Neural Network
Brief Title: Effects of ITBS Combined with NMES on Dysphagia After Stroke
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Luo Xiu, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-6-11
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Dysphagia; Intermittent Theta Burst Stimulation; Neuromuscular Electrical Stimulation; Functional Near-infrared Spectroscopy
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- iTBS combined with NMES (Experimental): On the basis of conventional treatment and swallowing rehabilitation training,The swallowing cortex of the affected hemisphere was stimulated with iTBS first, followed by NMES stimulation for 30 minutes after 10 minutes
  Interventions: Device: Transcranial magnetic stimulation
- iTBS combined with sham NMES (Experimental): On the basis of conventional treatment and swallowing rehabilitation training,The swallowing cortex of the affected hemisphere was stimulated with iTBS first, followed by NMES sham stimulation for 30 minutes after 10 minutes
  Interventions: Device: Transcranial magnetic stimulation
- sham iTBS combined with NMES (Experimental): On the basis of conventional treatment and swallowing rehabilitation training,The swallowing cortex of the affected hemisphere was stimulated with sham iTBS first, followed by NMES stimulation for 30 minutes after 10 minutes
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — The treatment parameter for iTBS was 80% stimulus intensity. The stimulation frequency was 50Hz in the plexus and 5Hz in the interplexus. Each burst stimulus consisted of 3 consecutive pulses, 2s stimulus, 8s interval, and repeated 20 times, a total of 600 pulses, and the duration of stimulation was 189s. NMES treatment parameters for output waveform for two-way square wave, wave width 700 ms, positive and negative half wave (300 ms) between 100 ms intermittent, stimulating frequency 50 hz, treatment when the output intensity range of 0 ~ 25 ma, stimulating electrodes pasted in bilateral mandibular hyoid muscle movement points, output intensity in patients with tongue bone muscle group it is advisable to have a sense of fashion, extrusion. Each treatment lasted 30 minutes, once a day, 5 times a week for 2 weeks.

SUMMARY:
In recent years, research on intermittent Theta Burst Stimulation (iTBS), as a special high-frequency （repetitive transcranial magnetic stimulation，rTMS） stimulation paradigm, has focused on exploring the effects in healthy people. Based on previous studies, it is believed that the central magnetic stimulation combined with peripheral electrical stimulation based on the "central-peripheral-central" closed-loop rehabilitation concept has the best effect, but there are few clinical studies on the efficacy and mechanism of iTBS combined treatment of dysphagia after stroke, and the selection of the optimal stimulation scheme and target has not yet been determined, therefore, this study aims to observe the efficacy and mechanism of implementation of iTBS combined with neuromuscular electrical stimulation (NMES) on with patients with dysphagia (PSD) .

DETAILED DESCRIPTION:
The purpose of this study is to observe the effect of intermittent Theta Burst Stimulation (iTBS) combined with neuromuscular electrical stimulation (NMES) on patients with dysphagia (PSD) after stroke, and to detect the activation of related swallowing networks in patients with PSD after receiving iTBS combined with NMES by functional near-infrared spectroscopy (fNIRS), and to explore the possible mechanism of PSD treatment, so as to provide a theoretical basis for finding the best, specific and individualized treatment plan for the treatment of PSD patients. Promote the functional recovery of patients, reduce complications, and promote the prognosis of diseases.

Patients who withdrew treatment for any reason other than progression (other than withdrawal of consent or loss to follow-up) continued to undergo objective assessment every 8 weeks to collect information on disease progression. Investigators were required to collect long-term follow-up information on survival by telephone at least every 12 weeks after documentation of disease progression by contacting patients, family members, or the patient's current treating physician.

Subjects who have the right to withdraw from the trial in the middle of the trial, or who are no longer tested and are lost to follow-up even though they have not explicitly proposed to withdraw from the trial, are also considered "withdrawal" (or "dropout"). The reasons for their withdrawal should be known as much as possible and documented. If the withdrawal is due to an adverse event, the patient should be visited for examination until the pre-treatment status or no clinical significance, and the adverse event form should be completed. The cause of the absconted case should be recorded in detail, and the informed consent form, original medical record, and case report form should be retained for future reference.

Treatment of drop-off cases: (1) When the subject falls off, the investigator should contact the subject to inquire about the reason as much as possible by visiting the door to make an appointment by telephone or letter. (2) If the experimental case is withdrawn due to allergic reactions, adverse reactions, or ineffective treatment, the investigator shall take corresponding treatment measures according to the actual situation of the subject. (3) The investigator should fill in the record of the main reason for discontinuing the trial. (4) All patients who have been selected and have been numbered, regardless of whether they have dropped out or not, should be recorded and kept for observation, both for filing and for intention-to-intention analysis (ITT), and all shedding cases should be summarized and statistically analyzed.

The sample size was calculated using G-power software based on the references.SPSS software was used for statistical description and analysis. Count data were expressed as rates or percentages, and chi-square tests were used for comparisons between groups. If the data conform to the normal distribution and the variance is homogeneous, (x̅ ± s) is used to express the continuous data, the one-way ANOVA was used for comparison between multiple groups, the least-significant difference (LSD) method was used for subsequent pairwise comparisons, and the paired sample t-test was used for comparison before and after treatment within the group. If the normal distribution is not conformed, the median and quartile M(P25,P75) are used, and the rank sum test is used. A P value of less than 0.05 indicated that the difference was statistically significant. The task state data processing of （functional near-infrared spectroscopy，fNIRS） is run by NirSpark toolkit software for data preprocessing. is run by NirSpark toolkit software for data preprocessing.

ELIGIBILITY:
Inclusion Criteria:

* 18 ~80 years old;
* The patients met the diagnostic criteria of stroke in the "Diagnostic Points for Major Cerebrovascular Diseases in China 2019" formulated by the Chinese Society of Neurology, and were confirmed by head CT or MRI;
* The patients met the diagnostic criteria of dysphagia in the "Chinese Expert Consensus on the Evaluation and treatment of Dysphagia (2017 edition)" and were confirmed by VFSS;
* The disease duration ranged from 2 weeks to 6 months;
* The vital signs of the patient were stable;
* The score of mini-mental state examination (MMSE) was more than 17 points for the illiterate, more than 20 points for the primary scholar, and more than 24 points for the secondary school or above;
* Can independently or under the auxiliary balance the seat 30 minutes or more;
* The skull was intact without craniotomy and/or cranioplasty;
* Informed consent was obtained from all subjects or their families.

Exclusion Criteria:

* A history of other diseases that may cause dysphagia, such as Parkinson's disease, head and neck radiotherapy, or other neurological diseases;
* Contraindications to iTBS or NMES with a history of epilepsy, intracranial metal implants, bleeding tendency, etc.;
* Skin damage and infection on the front of the neck affect the placement of the surface electrode;
* Such as fever, important viscera function failure condition is not stable, or critically ill.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
functional near-infrared spectroscopy | immediately before and immediately after the intervention
  Functional near-infrared spectroscopy (fNIRS) is a non-invasive neuroimaging technology based on blood vessels, which can be used to evaluate the activation of brain regions associated with swallowing
Standardized Swallowing Assessment Scale | immediately before and immediately after the intervention
  The Standard Swallowing Assessment Scale is a method of assessing a patient's swallowing function. During the assessment, the patient's level of consciousness, head and trunk control, breathing patterns, lip closure, soft palate movements, laryngeal function, gag reflex, and voluntary cough should be recorded.The highest score on the scale is 46 points, and the lowest score is 18 points, and the lower the score, the better the swallowing function.
The Yale Pharyngeal Residue Severity Rating Scale | immediately before and immediately after the intervention
  The Yale Pharyngeal Residue Severity Rating Scale is a laryngoscopy-based assessment scale used to assess the degree of food residue.The scale divided the residues of the valley of the eglottis and the piriform fossa into grades 1-5 according to the severity of the scale, respectively. The higher the grade, the more severe the food residue

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No